CLINICAL TRIAL: NCT00746642
Title: Use of Mellitor Sensor for Continuous Glucose Monitoring - An Ex-Vivo Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mellitor (Industry)
Responsible Party: Dr. Hanna Levy - study director, Melitor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MS-EV -1.0
Record Dates: First submitted 2008-09-03; First posted 2008-09-04 (Estimated); Last update posted 2009-06-04 (Estimated); Status verified 2009-06

CONDITIONS: Diabetes Mellitus
Keywords: glucose measurements
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Glucose measurements using "Mellitor" device.
  Interventions: Device: Mellitor device for glucose measurement
- B (Active Comparator): Glucose measurements conducted by using gold standard, "Yellow Springs" glucose analyzer
  Interventions: Device: Mellitor device for glucose measurement

INTERVENTIONS:
Device: Mellitor device for glucose measurement — Glucose measurement using "Mellitor" device

SUMMARY:
Most patients with diabetes mellitus have to measure their blood glucose levels quite often, in order to maintain a proper glycemic control. Current methods of self-monitoring of blood glucose are invasive, painful, uncomfortable, and only allow occasional, from time-to-time, measurements. Real-time continuous monitoring would provide a helpful tool for improvement of glycemic control, thus decreasing the incidence of hypoglycemia and improving glucose control. The Mellitor sensor is a new concept of continue glucose monitoring device. The Mellitor device is an implantable continuous glucose monitoring sensor that is intended for detection episodes of hyperglycemia and hypoglycemia in diabetic patients, and facilitates both acute and long-term therapy adjustments. This study was design in order to evaluate glucose measurement capabilities by the Mellitor sensor that is being developed. Transudate liquid samples, withdrawn in a clinical procedure and normally immediately disposed, will be used for glucose measurement by the Mellitor sensor.

Study Design

This study is an ex-vivo comparative study. 20 patients will be recruited for the study, according to patients' inflow and meeting eligibility criteria.

Study Goal

Study objective is to evaluate the feasibility of the Mellitor Sensor technology for glucose level measurement.

Study Endpoint

Mellitor technology feasibility will be established by comparing Mellitor glucose measurements results, based on transudate/exudates liquid withdrawal for other medical reasons, to "gold standard, Yellow Springs" glucose analyzer, or a comparable, calibrated and approved device using the same transudate/exudates liquid. Interdevice variability should be within 10%.

ELIGIBILITY:
Inclusion Criteria:

* Male/Female aged 18 and up.
* Subject was scheduled for transudate/exudate liquid withdrawal.
* Subject able to comprehend and give informed consent for participation in this study.
* Signed Informed Consent Form

Exclusion Criteria:

* Known cognitive or psychiatric disorder.
* Subjects with HIV.
* Subject refuses to sign inform consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-05 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
Mellitor technology feasibility will be established by comparing Mellitor glucose measurements results to "gold standard, Yellow Springs" glucose analyzer, or a comparable. Interdevice variability should be within 10%. | during glucose measurements

CONTACTS AND LOCATIONS:
Overall Officials: Roi Eldor, MD, Principal Investigator — Hadassah Medical Organization, Jerusalem
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel